CLINICAL TRIAL: NCT07353788
Title: Postoperative Complications and Outcomes Related to Mechanical Power in One-lung Ventilation- A Multicentre Observational Study
Brief Title: Mechanical Power in One-lung Ventilation
Acronym: POWEROL
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Clinical professor, Ankara University
Other Study IDs: 15.10.2025
Record Dates: First submitted 2025-12-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Thoracic Anesthesia; Thoracotomy Surgery
Keywords: one lung ventilation; mechanical power; postoperative pulmonary complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thoracic surgery usually necessitates one-lung ventilation (OLV) to provide surgical access while maintaining adequate gas exchange. However, OLV is associated with an increased risk of PPCs , a major cause of morbidity and mortality. Mechanical power, a composite parameter incorporating tidal volume, respiratory rate, driving pressure, and flow resistance, has been proposed as a key factor influencing ventilator-induced lung injury (VILI) and postoperative outcome. Understanding the association between mechanical power during OLV and PPCs could provide insights for optimizing intraoperative ventilatory strategies and reducing the burden of PPCs. As OLV inherently alters normal lung mechanics by decreasing functional residual capacity and introducing inequalities in ventilation-perfusion ratio, the complexity of managing mechanical power becomes even more pronounced. Under these altered conditions, the risk of PPC-including atelectasis, pneumonia, and respiratory failure-can be significantly elevated. Factors such as ventilatory settings, lung protection strategies, and the duration of OLV play pivotal roles in influencing mechanical power delivery and thereby impacting lung function recovery post-surgery. Current literature indicates a correlation between inappropriate mechanical ventilation strategies during OLV and increased incidence of PPCs. However, there remains a gap in understanding how precisely mechanical power, as a quantifiable measure, influences patient outcomes following OLV. Therefore, this study aims to investigate the relationship between mechanical power during OLV and the subsequent risk of PPC. By elucidating these dynamics, the findings may inform clinical practices surrounding OLV management, ultimately improving patient safety and outcomes in thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older,
2. ASA physical status I-IV
3. All thoracic surgeries
4. One lung ventilation period >1 hour
5. Patients capable of giving written informed consent

Exclusion Criteria:

1-Patients undergoing cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of PPCs during the first five postoperative days, defined according to standard criteria | From enrollment to the end of postoperative 5 th day
  Postoperative pulmonary complications ;(e.g., pneumonia, acute respiratory distress syndrome [ARDS], or prolonged mechanical ventilation).According to StEP-COMPAC group definition [Abbott et al. 2018 Br J Anaesth 2018 May;120(5):1066-1079.]

SECONDARY OUTCOMES:
Threshold mechanical power (J/min)associated with PPCs | From enrollment to postoperative 5 th day
Unscheduled ICU admission rates | From enrollment to postoperative 5 th day
Extra-pulmonary postoperative complications(number of complications) | From enrollment to postoperative 5 th day
Length of ICU stay(day) | up to 5 th day
Length of hospital stay(day) | From enrollment to postoperative 5 th day

IPD SHARING:
Plan to Share IPD: Undecided